CLINICAL TRIAL: NCT03412357
Title: MesoTRAP: A Pilot Clinical Trial and Feasibility Study Comparing Video-assisted Thoracoscopic Partial Pleurectomy/Decortication With Indwelling Pleural Catheter in Patients With Trapped Lung Due to Malignant Pleural Mesothelioma Designed to Address Recruitment and Randomisation Uncertainties and Sample Size Requirements for a Phase III Trial.
Brief Title: MesoTRAP: A Study Comparing Video-assisted Thoracoscopic Partial Pleurectomy/Decortication With Indwelling Pleural Catheter in Patients With Trapped Lung Due to Malignant Pleural Mesothelioma.
Acronym: MesoTRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); London School of Hygiene and Tropical Medicine (Other); King's College London (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO2128
Record Dates: First submitted 2017-11-29; First posted 2018-01-26 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Malignant Pleural Mesothelioma; Trapped Lung
Keywords: pleurectomy/decortication; indwelling pleural catheter
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cerebral Decortication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pleurectomy/decortication (Experimental)
  Interventions: Procedure: pleurectomy/decortication
- indwelling pleural catheter (Experimental)
  Interventions: Procedure: indwelling pleural catheter

INTERVENTIONS:
Procedure: pleurectomy/decortication — VAT-PD is a type of "keyhole surgery" performed under general anaesthesia using a telescope and instruments put inside the chest. Through small incisions, or keyholes made between the ribs, the thoracic surgeon removes the hard rind of the tumour over the surface of the lung, thereby allowing the 'trapped' lung to fully expand again. Simultaneous removal of mesothelioma from the outer pleural membrane allows pleurodesis to occur.
  Other Names: video-assisted thoracoscopic partial pleurectomy/decortication; VAT-PD
  Arms: pleurectomy/decortication
Procedure: indwelling pleural catheter — A soft silicone catheter (IPC) with a one-way valve at the end is inserted a few centimetres under the skin under local anaesthesia. The inside end of the catheter is inserted into the pleural space and the outside end is connected to a vacuum drainage bottle. The IPC permits regular fluid drainage.
  Other Names: IPC
  Arms: indwelling pleural catheter

SUMMARY:
Malignant pleural mesothelioma is a cancer, caused by asbestos, which currently affects 2500 people in the UK each year. The main symptom is breathlessness caused by fluid building up in the space between the lung and the chest wall (pleural effusion). Treatment involves draining the fluid to allow the lung to re-expand (pleurodesis). However, sometimes tumour growth over the surface of the lung can prevent it from re-expanding. This 'trapped' lung results in fluid re-accumulation and repeated drainage which can lead to discomfort and multiple hospital visits.

One approach to dealing with 'trapped' lung in mesothelioma is to insert a thin tube (Indwelling Pleural Catheter - IPC) into the space around the lung. The tube can stay in place for a long time allowing patients to drain off fluid at home.

Another approach is a keyhole surgical operation (video-assisted thoracoscopic partial pleurectomy/decortication - VAT-PD) to remove as much tumour as possible from the lining of the lung to allow it to re-expand.

While both approaches are currently offered in clinical practice, it is not known which of the two is most effective at relieving breathlessness. The only way to find out is to conduct a research trial comparing the two. The Investigators plan to do this, but first of all need to carry out a small pilot study to collect information necessary to help plan the full study.

DETAILED DESCRIPTION:
This is a multi-centre, open-label, randomised controlled pilot clinical trial and feasibility study comparing video-assisted thoracoscopic partial pleurectomy/decortication (VAT-PD) with indwelling pleural catheter (IPC) in patients with trapped lung (TL) and pleural effusion due to malignant pleural mesothelioma (MPM), aimed at addressing recruitment and randomisation uncertainties as well as sample size requirements for a full phase III study. 38 patients will be randomised and allocated in a 1:1 ratio to either VAT-PD or IPC.

The study will be undertaken at mesothelioma surgical centres with expertise in either IPC, VAT-PD or both procedures, together with their linked non-surgical referral hospitals (hub and spoke). Patients meeting all eligibility criteria will be informed about the study, provided with a patient information sheet and given at least 24 hours to consider participation.

Following consent, patients will be randomised, baseline measurements will be taken and a procedure date will be arranged. Following the procedure follow-up visits at 6 weeks, 3, 6 and 12 months post-randomisation are planned to coincide with clinical care visits.

In parallel with the main study an observational sub-study will collect observational data on a cohort of patients who have Malignant Pleural Mesothelioma and trapped lung, but who are either not eligible to participate, or who decline to participate in the main study. Patients in the Observational Sub-study will receive the same baseline and follow-up visits as those in the main study, but will receive standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed MPM
2. Trapped lung, defined as a 'clinically significant trapped lung requiring intervention in the opinion of the clinical team"
3. Pleural effusion present (following re-accumulation)
4. Considered by the clinical team to be suitable and fit enough to undergo VAT-PD
5. Community services or patient/carer able to drain IPC at least twice weekly
6. Considered by the clinical team to be equally suitable for treatment with VAT-PD or IPC, and therefore eligible for treatment allocation by randomisation.
7. Patient willing to receive either VAT-PD or IPC and attend the respective designated centre for their treatment
8. Expected survival of at least 4 months, as assessed by managing clinician
9. Age ≥ 18 years
10. Able to provide informed consent

Exclusion Criteria:

1. Lung re-expands fully following pleural fluid drainage i.e. no entrapment
2. Evidence of active pleural infection
3. Current participation in an RCT or CTIMP
4. Females: pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
To measure the standard deviation of Visual Analogue Scale scores for breathlessness | Daily from randomisation to 12 months
  The Visual Analogue Scale (VAS) is a 100mm line for patients to record the severity of a their breathlessness where 0mm is "No breathlessness at all" and 100mm is "Worst possible breathlessness".

SECONDARY OUTCOMES:
To measure the standard deviation of Visual Analogue Scale scores for chest pain | Daily from randomisation to 12 months
  The Visual Analogue Scale (VAS) is a 100mm line for patients to record the severity of a their chest pain where 0mm is "No pain at all" and 100mm is "Worst possible pain".
Quality of Life measured using the EQ-5D-5L | Baseline, intervention, 6 weeks, 3, 6 and 12 months post randomisation
Quality of Life measured using the EORTC QLQC30 | Baseline, intervention, 6 weeks, 3, 6 and 12 months post randomisation
Survival at 30 days and 12 months post randomisation | 30 days and 12 months post randomisation
Adverse events | From randomisation to the end of study follow-up (expected to be 12 months)
The prevalence of trapped lung in patients with MPM | From beginning to end of recruitment period (18 months)
Percentage of eligible patients in participating centres | From beginning to end of recruitment period (18 months)
Recruitment rate | From beginning to end of recruitment period (18 months)
To assess completion of resource use data during follow-up using patients' routine data | Baseline, intervention, 6 weeks, 3, 6 and 12 months post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rintoul, Dr, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (18):
- United Kingdom (18):
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - North Bristol NHS Trust, Bristol
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Cambridge University Hospitals, Cambridge
  - Derby Teaching Hospitals NHS Foundation Trust, Derby
  - Golden Jubilee National Hospital, Glasgow
  - Queen Elizabeth University Hospital and New Victoria Hospital, Glasgow
  - University Hospitals of Leicester, Leicester
  - Barts Health NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Pennine Acute Hospitals NHS Trust, Manchester
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Sheffield Teaching Hospitals, Sheffield
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

REFERENCES:
- [Derived] Matthews C, Freeman C, Sharples LD, Fox-Rushby J, Tod A, Maskell NA, Edwards JG, Coonar AS, Sivasothy P, Hughes V, Rahman NM, Waller DA, Rintoul RC. MesoTRAP: a feasibility study that includes a pilot clinical trial comparing video-assisted thoracoscopic partial pleurectomy decortication with indwelling pleural catheter in patients with trapped lung due to malignant pleural mesothelioma designed to address recruitment and randomisation uncertainties and sample size requirements for a phase III trial. BMJ Open Respir Res. 2019 Jan 5;6(1):e000368. doi: 10.1136/bmjresp-2018-000368. eCollection 2019. PMID 30687504